CLINICAL TRIAL: NCT00256113
Title: An Eight-Week, Multicenter, Double-blind, Placebo-controlled Study Evaluating the Efficacy, Safety, and Tolerability of One Fixed 100 mg Dose of Saredutant in Patients With Major Depressive Disorder
Brief Title: An Eight-week Study to Evaluate the Efficacy and Safety of Saredutant in Patients With Depression
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EFC5575
Record Dates: First submitted 2005-11-07; First posted 2005-11-21 (Estimated); Last update posted 2018-04-20 (Actual); Status verified 2018-04

CONDITIONS: Depressive Disorder
Keywords: depression; antidepressive agents; controlled clinical trial
MeSH Terms: conditions — Depressive Disorder; Depression | interventions — SR 48968

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: Saredutant succinate (SR48968C)

SUMMARY:
The purpose of the study is to evaluate the efficacy and safety of saredutant (or SR48968C) in patients with depression.

The primary objective is to evaluate the efficacy of a 100 mg dose of saredutant compared to placebo in patients with depression.

The secondary objectives are to evaluate the safety of saredutant, to evaluate the efficacy of saredutant on disability and quality of life in patients with depression, and to evaluate blood levels of saredutant.

DETAILED DESCRIPTION:
The study is a multicenter, multicountry, randomized, parallel-group, double blind, placebo and paroxetine-controlled study consisting of three segments (A, B, and C). Segment A is a 1-week, placebo, single-blind period and Segment B is an 8-week, double blind period. Patients completing Segment B may be eligible for enrollment into Segment C, a 44-week, double blind extension. All randomized patients must complete a post-study visit 1 week after intake of the last dose of study medication.

ELIGIBILITY:
Inclusion Criteria:

* 1. Male or female patients.
* 2. 18 to 64 years of age.
* 3. Inpatients or outpatients.
* 4. Written informed consent from the patient and/or legally authorized representative.
* 5. Able to comply with the protocol and follow written and verbal instructions.
* 6. Subjects of childbearing potential must have a confirmed negative serum b-hCG test prior to entry into Segment B and must employ an acceptable method of birth control (e.g., oral, depot, or implanted contraceptive method, IUDs, sterilization, barrier methods in conjunction with spermicide).
* 7. Diagnosis of major depressive disorder, as defined by Diagnostic and Statistical Manual of Mental Disorders, 4th edition, Text Revision criteria and confirmed by the semi-structured Mini International Neuropsychiatric Interview (MINI), recurrent episode for at least one month prior to the entry.
* 8. Minimum total score of 22 on the Montgomery-Asberg Depression Rating Scale (MADRS).

Exclusion Criteria:

* 1. Patients whose current depressive episode is diagnosed with psychotic features, catatonic features, seasonal pattern or post-partum onset.
* 2. The duration of the current depressive episode is greater than 2 years.
* 3. Patients who are currently suicidal or have a history of a suicide attempt within 3 years prior to entry.
* 4. Patients whose current depressive episode is secondary to a general medical disorder.
* 5. Patients with a history or presence of bipolar disorders or psychotic disorders according to the D and L criteria of the MINI.
* 6. Patients with alcohol dependence or abuse or substance dependence or abuse in the past 12 months except nicotine or caffeine dependence.
* 7. Patients with a history of failure to respond to treatment with paroxetine or other antidepressant medications.*
* 8. Patients who have used the following prior to entry into Segment B: any antipsychotic within 3 months,-fluoxetine within 35 days, -any monoamine oxidase inhibitor within 21 days, any other antidepressant, anxiolytic, sedative-hypnotic, or mood-stabilizer (lithium, anticonvulsants) within 7 days except permitted concomitant medications.
* 9. Females who are pregnant or breast-feeding.
* 10. Severe or unstable cardiovascular, renal, hepatic, respiratory, hematological, endocrinological, neurological, or other somatic disease that might interfere with the evaluation of study medication.
* 11. History of seizures other than a single childhood febrile seizure.
* 12. ECG abnormalities of potential clinical significance including a QT interval with Bazett's correction of 500 msec or more at entry.
* 13. Use of known inducers or potent inhibitors of CYP3A4 within 7 days of entry.
* 14. Use of drugs with known risk for Torsade de Pointes within 7 days of entry into Segment B.
* 15. Participation in a clinical trial of an experimental therapy within 30 days prior to entry or prior participation in a clinical trial of saredutant.
* 16. Patients with a positive HbsAg or anti-HCV antibody test at screening.
* 17. Patients with any of the following at screening: ALT >2 times the upper limit of the normal range (XULN), AST >2XULN, GGT >3XULN, total or conjugated bilirubin >ULN

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 467 (Actual)
Dates: Start 2004-12; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
The primary outcome of the study is the change from baseline to Day 56 of treatment in the Hamilton Depression Rating Scale (HAM-D) total score.

SECONDARY OUTCOMES:
The main secondary outcomes are the changes from baseline to Day 56 of treatment in the HAM-D depressed mood item, the Montgomery Asberg Depression Rating Scale total, and the Clinical Global Impression Severity of Illness scores.

CONTACTS AND LOCATIONS:
Overall Officials: ICD CSD, Study Director — Sanofi
Locations (8):
- Sanofi-Aventis Administrative Office, Laval, Canada
- Sanofi-Aventis Administrative Office, Santiago, Chile
- Sanofi-Aventis Administrative Office, Zagreb, Croatia
- Sanofi-Aventis Administrative Office, Prague, Czechia
- Sanofi-Aventis Administrative Office, Tallinn, Estonia
- Sanofi-Aventis Administrative Office, Berlin, Germany
- Sanofi-Aventis Administrative Office, México, Mexico
- Sanofi-Aventis Administrative Office, Porto Salvo, Portugal

REFERENCES:
- See also: Related Info — http://www.sanofi-aventis.com